CLINICAL TRIAL: NCT07108738
Title: Exploring Natural Alternatives: Pomegranate Peel Extract for Primary Molar Pulpotomy
Brief Title: Pomegranate Peel Extract for Primary Molar Pulpotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, associate professor of pediatric dentistry, faculty of dentistry, Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #R-PED-7-25-3206
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Pulpitis Reversible; Pulp Exposure, Dental
Keywords: Pulpotomy; Primary molars; Pomegranate Peel Extract; Mineral Trioxide Aggregate
MeSH Terms: conditions — Dental Pulp Exposure | interventions — Pulpotomy; Radiation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: zinc oxide-pomegranate peel extract paste (Experimental): 30 primary molars will be treated with pomegranate peel extract freshly mixed with zinc oxide powder till it reaches a suitable consistency (1:1 ratio by volume) to cover pulp stumps
  Interventions: Procedure: Pulpotomy; Procedure: Radiation
- group 2: MTA (Active Comparator): 30 primary molars will be treated with MTA to cover pulp stumps
  Interventions: Procedure: Pulpotomy; Procedure: Radiation

INTERVENTIONS:
Procedure: Pulpotomy — Teeth will be anesthetized then Rubber dam and high suction will be used in pulpotomy procedure. Cavity outline will be performed by sterile #330 high speed bur using water spray. Caries will be removed by large spoon excavator. When pulpal exposure occurred, the roof of pulp chamber will be removed by low speed round bur. Haemostasis will be obtained by applying pressure with a moist cotton pellet with saline. Then the test materials will be applied. after that, pulp stumps of all molars in each group will be dressed using Intermediate restorative material, then the tooth will be restored with a preformed stainless steel crown
Procedure: Radiation — Radiographic evaluation will be performed immediately after teeth restoration (baseline radiograph), then after three, six, and twelve months for the furcation radiolucency area and bone radiodensity. A photo-simulated phosphorus plate sensor was used to take direct standardized digital radiographs. The parallel periapical technique was obtained by Rinn, which is attached to the X-ray tube with its arm fastened to the film holder that contained a coated PSP (photo-stimulated phosphorus plate). To ensure standardization during radiographic film retakes, condensation rubber base impression material will be positioned on the outside of the film holder, and the child is told to bite on it while the material is set. The sensor wil exposed to an X-ray machine (Planmeca ProX, Helsinki, Finland) with a central ray perpendicular to the sensor at 70 kVp, 6 mA, and 0.8 s. Radio-densitometric and radiometric analysis of the radiographs will be performed by RadiAnt software.

SUMMARY:
Pomegranate peel extract has demonstrated a range of potential uses in the biomedical industry in recent years because of its numerous benefits, which include anti-inflammatory, antibacterial, anti-apoptotic, antioxidant, and cell-regeneration-promoting qualities. Therefore, the purpose of this study will be to evaluate the clinical and radiographic efficacy of Pomegranate peel extract as a pulpotomy agent in primary teeth.

DETAILED DESCRIPTION:
A total of sixty primary molars in thirty children aged between 4 and 8 years will be randomly divided into two groups: Group I, the Pomegranate peel extract group, and Group II, the MTA group. After pulpotomy treatment, all molars will be restored with stainless steel crowns. Follow-up will be done after 3, 6, and 9 months for clinical and radiographic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Restorable primary molars with deep carious lesions.
* Absence of gingival swelling or sinus tract.
* Absence of spontaneous pain
* Absence of pain on percussion.
* Absence of discontinuity of lamina dura
* Absence of internal root resorption.
* Absence of external root resorption.
* Absence of inter-radicular or periapical bone destruction (radiolucency).

Exclusion Criteria:

* presence of spontaneous pain
* presence of gingival swelling or sinus tract
* presence of internal or external root resorption
* pain on percussion.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
absence of pain | up to 9 months
  Measuring Method: Verbal Question to Patient /Parents Measuring Unite: score 0 for absence of pain and score 1 for presence of pain
absence of fistula | up to 9 months]
  Measuring Method: Visual examination by operator Measuring Unit: score 0 for absence of swelling and score 1 for presence of swelling
Tenderness to percussion | up to 9 months
  Measuring Method: Percussion test Measuring Unite: Binary (+/-)
Furcation radiolucency | 3 months
  Measuring Method: periapical x-ray for assessment of radio-density of bone at the furcation area, Measuring Unit: mean value of gray level (which measures density scale between 0 to 256, with zero being the lowest value and 256 the highest dense value)
furcation radiolucency | 6 months
  Measuring Method: periapical x-ray for assessment of radio-density of bone at the furcation area, Measuring Unit: mean value of gray level (which measures density scale between 0 to 256, with zero being the lowest value and 256 the highest dense value)
furcation radiolucency | 9 months
  Description: Measuring Method: periapical x-ray for assessment of radio-density of bone at the furcation area, Measuring Unit: mean value of gray level (which measures density scale between 0 to 256, with zero being the lowest value and 256 the highest dense value)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

REFERENCES:
- [Background] Mushtaq A, Nangia T, Goswami M. Comparative Evaluation of the Treatment Outcomes of Pulpotomy in Primary Molars Using Mineral Trioxide Aggregate and 3Mixtatin: A Randomized Clinical Trial. Int J Clin Pediatr Dent. 2023 Nov-Dec;16(6):810-815. doi: 10.5005/jp-journals-10005-2720. PMID 38344366
- [Background] Farsi N, Alamoudi N, Balto K, Mushayt A. Success of mineral trioxide aggregate in pulpotomized primary molars. J Clin Pediatr Dent. 2005 Summer;29(4):307-11. doi: 10.17796/jcpd.29.4.n80t77w625118k73. PMID 16161395